CLINICAL TRIAL: NCT06765434
Title: The Effects of Personalized Music Listening on Functional and Cognitive Status in Advanced-Stage Alzheimer's Disease
Brief Title: Effects of Personalized Music Listening in Advanced Alzheimer's
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Emine Atıcı, Associate Professor, Okan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 013
Record Dates: First submitted 2025-01-03; First posted 2025-01-09 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer Disease, Late Onset; Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Experimental): The control group will listen to No. 2 from Dmitri Shostakovich's Jazz Waltz Suite played from a CD player for 12 weeks, 3 days per week.
  Interventions: Other: Music ( Dmitri Shostakovich's Jazz Waltz Suite)
- Personalized music (Experimental): In the experimental group, music that has created positive impacts in the participants' lives will be identified and played from a CD player for 12 weeks, 3 days per week.
  Interventions: Other: Music( Personalized music)

INTERVENTIONS:
Other: Music ( Dmitri Shostakovich's Jazz Waltz Suite) — Music
  Arms: Control
Other: Music( Personalized music) — Music
  Arms: Personalized music

SUMMARY:
Recent functional imaging studies have facilitated a better understanding of the neuroplasticity mechanisms underlying the strong and multifaceted effects of music on brain development. For this reason, music is considered a significant factor in improving recall and mood in individuals with dementia.

A review investigating the cognitive and behavioral effects of music listening in Alzheimer's disease (AD) reported that personalized (individualized) music listening yielded the best outcomes.

This study aims to examine the effects of personalized music activities on functional and cognitive status in individuals with advanced-stage AD.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 and over
* Patients diagnosed with advanced-stage Alzheimer's type dementia according to the diagnostic criteria of the American Psychiatric Association's Diagnostic and Statistical Manual of Mental Disorders (DSM-V)

Exclusion Criteria:

* Patients with hearing impairments that could interfere with music listening
* Individuals who have received music education and are able to play an instrument
* Patients with a history of heart disease, hypertension, or diabetes will be excluded from the study.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 54 (Actual)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Standardized Mini-Mental State Examination (SMMSE) | baseline and 12 week later
  First introduced in 1975 by Folstein and colleagues, this test is one of the most widely used tools for quantitatively assessing cognitive performance within standard europsychiatric examination methods. It was developed as a brief cognitive assessment tool. The test holds particular significance in evaluating elderly patients. Its validity and reliability have been confirmed in many countries. In Turkey, the validity and reliability study was conducted by Güngen and colleagues. Although it has limited specificity for distinguishing clinical syndromes, it is a short, practical, and standardized test suitable for assessing overall cognitive levels.
  The SMMSE evaluates cognitive functions across five domains: orientation, registration, attention and calculation, recall, and language. The total score is 30. Scores of 24 or below indicate the need for evaluation for dementia. The inter-rater reliability study reported an r-value of 0.99 and a kappa value of 0.92.
  Sample Questio
Functional Independence Measure (FIM) | baseline and 12 week later
  Developed by Hamilton et al. (1994), the scale measures the degree of independence in individuals' basic physical and cognitive functions in daily living activities. The FIM consists of 18 items and assesses two main domains: motor (13 items) and cognitive (5 items). The maximum scores for the Functional Independence Measure in motor (FIM-M) and cognitive (FIM-C) are 91 and 35, respectively. The total FIM score can range from 18 to 126. It includes six functional areas: self-care, sphincter control, mobility, locomotion, communication, and social perception. Each item is evaluated using a 7-point scale, and the total score is 126.
  The Turkish validity and reliability study for the scale was conducted by Küçükdeveci et al. in 2001. The internal consistency was found to be above 0.48 for individuals with spinal cord injuries and 0.44 for stroke patients.
Frontal Assessment Battery (FAB) | baseline and 12 week later
  The Frontal Assessment Battery, developed by Dubois et al., is a simple, easy-to-administer, and brief (approximately 10 minutes) bedside test designed to assess frontal lobe functions. It is useful in evaluating frontal lobe functions and detecting executive dysfunctions, as well as distinguishing degenerative diseases involving cortical-subcortical structures and monitoring the progression of these diseases. The FAB consists of 6 items, each scored on a 0-3 scale, with higher scores indicating better performance. The Turkish validity and reliability study was conducted by Güleç et al. (2009), and the internal consistency was found to be 0.65.
  The FAB consists of 6 subtests:
  Similarities (conceptualization) Word Fluency (mental flexibility) Motor Series (programming) Contradictory Instructions (sensitivity to interference) Action-Nonaction (inhibition control) Environmental Autonomy (capturing behavior)

SECONDARY OUTCOMES:
Clock Drawing Test (CDT) | baseline and 12 week later
  The Clock Drawing Test is an important tool for assessing cognitive parameters, specifically evaluating the ability to understand and plan, which are components of constructive praxis. The patient is asked to draw a clock, place the numbers on it, and mark the indicated time. It is scored on a scale of 6 points, with a score below 4 indicating impaired cognitive function.
  The scoring is as follows:
  Writing the number 12 in the correct position = 3 points Writing all 12 numbers = 1 point Drawing the hour and minute hands = 1 point Correctly marking the indicated time = 1 point. The Clock Drawing Test (CDT) is a simple neuropsychometric tool that can be easily applied to assess various neuropsychiatric functions. It was introduced by Critchley (1953) as an indicator of structural apraxia in the early 20th century. A Turkish norm and validity-reliability study of the CDT was conducted by Cangoz et al. in a population aged 50 and above.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Okan University, Istanbul, Turkey (Türkiye)